CLINICAL TRIAL: NCT00293592
Title: Dexamethasone for Cardiac Surgery Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, D van Dijk, Anesthesiologist/Intensivist, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DECS
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Systemic Inflammatory Response Syndrome; Cardiac Diseases; Postoperative Complications
Keywords: Heart surgery; Cardiopulmonary bypass; Systemic Inflammatory Response Syndrome (SIRS)
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Heart Diseases; Postoperative Complications | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 1 mg per kg as a single dose before initiation of cardiopulmonary bypass

SUMMARY:
This is a multicenter, randomized, double-blind trial, comparing clinical outcomes after the administration of high-dose dexamethasone versus placebo in patients undergoing heart surgery with the use of cardiopulmonary bypass. The primary endpoint is the occurrence of major complications (including all-cause mortality, myocardial infarction, stroke, renal failure, and prolonged mechanical ventilation) in the first 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All types of cardiac surgery in which cardiopulmonary bypass is used

Exclusion Criteria:

* Age under 18 years
* Life-expectancy < 6 months
* Emergency operations
* Re-operations within the same admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Actual)
Dates: Start 2006-05; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of mortality, myocardial infarction, stroke, renal failure and prolonged mechanical ventilation (> 48h) | 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: CJ Kalkman, MD, PhD, Study Chair — UMC Utrecht; D van Dijk, MD, PhD, Study Director — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Ottens TH, Hendrikse J, Slooter AJ, van Herwerden LA, Dieleman JM, van Dijk D. Low incidence of early postoperative cerebral edema after coronary artery bypass grafting. J Cardiothorac Vasc Anesth. 2015;29(3):632-6. doi: 10.1053/j.jvca.2014.12.004. Epub 2014 Dec 3. PMID 25817849
- [Result] van Osch D, Dieleman JM, van Dijk D, Jacob KA, Kluin J, Doevendans PA, Nathoe HM; DExamethasone for Cardiac Surgery (DECS) study group; DExamethasone for Cardiac Surgery DECS study group. Dexamethasone for the prevention of postoperative atrial fibrillation. Int J Cardiol. 2015 Mar 1;182:431-7. doi: 10.1016/j.ijcard.2014.12.094. Epub 2015 Jan 8. PMID 25596472
- [Result] Jacob KA, Dieleman JM, Nathoe HM, van Osch D, de Waal EE, Cramer MJ, Kluin J, van Dijk D. The effects of intraoperative dexamethasone on left atrial function and postoperative atrial fibrillation in cardiac surgical patients. Neth Heart J. 2015 Mar;23(3):168-73. doi: 10.1007/s12471-014-0638-5. PMID 25475514
- [Result] Ottens TH, Dieleman JM, Sauer AM, Peelen LM, Nierich AP, de Groot WJ, Nathoe HM, Buijsrogge MP, Kalkman CJ, van Dijk D; DExamethasone for Cardiac Surgery (DECS) Study Group. Effects of dexamethasone on cognitive decline after cardiac surgery: a randomized clinical trial. Anesthesiology. 2014 Sep;121(3):492-500. doi: 10.1097/ALN.0000000000000336. PMID 25225745
- [Result] Bunge JJ, van Osch D, Dieleman JM, Jacob KA, Kluin J, van Dijk D, Nathoe HM; Dexamethasone for Cardiac Surgery (DECS) Study Group. Dexamethasone for the prevention of postpericardiotomy syndrome: A DExamethasone for Cardiac Surgery substudy. Am Heart J. 2014 Jul;168(1):126-31.e1. doi: 10.1016/j.ahj.2014.03.017. Epub 2014 Apr 5. PMID 24952869
- [Result] Sauer AM, Slooter AJ, Veldhuijzen DS, van Eijk MM, Devlin JW, van Dijk D. Intraoperative dexamethasone and delirium after cardiac surgery: a randomized clinical trial. Anesth Analg. 2014 Nov;119(5):1046-52. doi: 10.1213/ANE.0000000000000248. PMID 24810262
- [Result] Dieleman JM, Nierich AP, Rosseel PM, van der Maaten JM, Hofland J, Diephuis JC, Schepp RM, Boer C, Moons KG, van Herwerden LA, Tijssen JG, Numan SC, Kalkman CJ, van Dijk D; Dexamethasone for Cardiac Surgery (DECS) Study Group. Intraoperative high-dose dexamethasone for cardiac surgery: a randomized controlled trial. JAMA. 2012 Nov 7;308(17):1761-7. doi: 10.1001/jama.2012.14144. PMID 23117776
- [Derived] Sauer AC, Veldhuijzen DS, Ottens TH, Slooter AJC, Kalkman CJ, van Dijk D. Association between delirium and cognitive change after cardiac surgery. Br J Anaesth. 2017 Aug 1;119(2):308-315. doi: 10.1093/bja/aex053. PMID 28854542
- [Derived] Jacob KA, Leaf DE, Dieleman JM, van Dijk D, Nierich AP, Rosseel PM, van der Maaten JM, Hofland J, Diephuis JC, de Lange F, Boer C, Kluin J, Waikar SS; Dexamethasone for Cardiac Surgery (DECS) Study Group. Intraoperative High-Dose Dexamethasone and Severe AKI after Cardiac Surgery. J Am Soc Nephrol. 2015 Dec;26(12):2947-51. doi: 10.1681/ASN.2014080840. Epub 2015 May 7. PMID 25952257
- [Derived] Ottens TH, Nijsten MW, Hofland J, Dieleman JM, Hoekstra M, van Dijk D, van der Maaten JM. Effect of high-dose dexamethasone on perioperative lactate levels and glucose control: a randomized controlled trial. Crit Care. 2015 Feb 13;19(1):41. doi: 10.1186/s13054-015-0736-9. PMID 25886901